CLINICAL TRIAL: NCT05072925
Title: Abuse Liability and Puffing Topography Assessments of the BIDI Stick Electronic Nicotine Delivery System (ENDS) in Comparison to a Combustible Cigarette and JUUL Pod-Based ENDS
Brief Title: BIDI Stick ENDS Abuse Liability and Puffing Topography Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BIDI Vapor (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BIDI-PK-01
Record Dates: First submitted 2021-09-26; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: E-cigarette Use; Cigarette Smoking
MeSH Terms: conditions — Vaping; Cigarette Smoking | interventions — Tobacco Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Combustible Cigarette (Active Comparator): The usual brand of combustible cigarette smoked by study subjects, with a minimum Federal Trade Commission tar yield of 8mg
  Interventions: Other: Tobacco products
- BIDI Stick ENDS Arctic flavor (Experimental): BIDI Stick ENDS containing 6% nicotine and Arctic flavor
  Interventions: Other: Tobacco products
- BIDI Stick ENDS Classic flavor (Experimental): BIDI Stick ENDS containing 6% nicotine and Classic flavor
  Interventions: Other: Tobacco products
- BIDI Stick ENDS Zest flavor (Experimental): BIDI Stick ENDS containing 6% nicotine and Zest flavor
  Interventions: Other: Tobacco products
- BIDI Stick ENDS Regal flavour (Experimental): BIDI Stick ENDS containing 6% nicotine and Regal flavor
  Interventions: Other: Tobacco products
- BIDI Stick ENDS Winter flavour (Experimental): BIDI Stick ENDS containing 6% nicotine and Winter flavor
  Interventions: Other: Tobacco products
- BIDI Stick ENDS Solar flavor (Experimental): BIDI Stick ENDS containing 6% nicotine and Solar flavor
  Interventions: Other: Tobacco products
- JUUL ENDS Virginia Tobacco flavor (Active Comparator): JUUL ENDS containing 5% nicotine and Virginia Tobacco flavor
  Interventions: Other: Tobacco products

INTERVENTIONS:
Other: Tobacco products — Products will be used under defined (10 puffs, 30 seconds apart) and ad libitum puffing conditions

SUMMARY:
This study assessed the abuse liability (measured by assessing how much nicotine enters the body when the BIDI Stick is used, and how this makes users feel) and puffing topography (puff characteristics like volume and duration) of the BIDI Stick ENDS, a type of electronic cigarette.

DETAILED DESCRIPTION:
This is a part-randomized, open label abuse liability assessment (ALA) and puffing topography study of nicotine-containing products carried out in 18 healthy adult volunteers who smoke combustible cigarettes.

Subjects will attend the study site 8 times (Visits 2-9) during the main study for ALA and puff topography assessments. Prior to each visit, subjects will be required to refrain from using any nicotine-containing products for a period of at least 12 hours before study product use.

At Visit 2, the subjects will smoke their usual brand cigarette during 2 use sessions. In the first session, subjects will smoke a single combustible cigarette of their usual brand by taking 10 puffs, 30 seconds apart. Blood samples will be obtained for plasma nicotine analysis, and blood pressure and heart rate will be recorded. Subjects will be asked to complete subjective effects questionnaires at various points either before, during, or after product use.

In the second session, which will begin immediately after the last blood draw following the first session and after all questionnaires have been completed, subjects will be allowed to take ad libitum puffs on their usual brand cigarette for a period of 60 minutes (1 hour). In a randomly-selected subset of 8 subjects, during this ad libitum puffing session puffing topography measurements will be made with a CReSS Pocket device. Subjects may smoke as many cigarettes as they like. In all subjects, a blood sample for nicotine PK analysis will be drawn at the end of the session. Blood pressure and heart rate will be recorded at this time. Subjective effects questionnaires will also be completed at specified timepoints.

At Visits 3-9, the subjects will use their randomly-assigned ENDS product during 2 use sessions. These use sessions, and the assessments made, will be the same as at visit 2. Prior to visit 3-9, subjects will be provided with a supply of their randomly-assigned product to use at home before their next visit (familiarization). This familiarization period should last a minimum of 2 and a maximum of 5 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females within the ages of 21 to 65 years, inclusive.
2. Subjects will have a body mass index (BMI) of 18.5 to 35.0 kg/m2, inclusive, and a body weight exceeding 52 kg (males) or 45 kg (females).
3. Subjects must be current smokers (≥10 per day) of factory-made, high tar (10mg) combustible cigarettes (eCO >10 ppm at screening) for at least one continuous year before Visit 1 and may be occasional or dual users of e-cigarettes.
4. Urine cotinine >200 ng/mL.
5. Subject demonstrates understanding of the study and willingness/consent to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the consent form.
6. Subject understands and is willing, able, and likely to comply with all the study procedures and restrictions.
7. Subject is in good general health in the opinion of the investigator, with no clinically significant and relevant abnormalities of medical history (e.g., uncontrolled hypertension, recent myocardial infarction or unstable angina, history of seizures or recent stomach ulcer).
8. Subject has a seated systolic blood pressure ≤160 mmHg, diastolic blood pressure ≤95 mmHg, and heart rate ≤100 bpm.
9. Females of childbearing potential are, in the opinion of the investigator, practicing a reliable method of contraception.

Exclusion Criteria:

1. Subjects who, in the judgment of the study physician, have recent or active COVID 19 infection, as evidenced by the following:

   1. Endorsement of symptoms that could indicate COVID-19 during screening (Section 13.1) and/or
   2. Body temperature ≥38.0°C and/or
   3. Laboratory test results suggestive of active or recent exposure to SARS-CoV-2 (Section 9.4).
2. Laboratory serology results positive for HBsAg, hepatitis C virus (HCV) antibody, (HIV) type 1 or 2.
3. Subjects who have participated in another clinical study within 30 days of Visit 1 or who have previously participated in this study.
4. Subjects who have an acute illness (e.g., upper respiratory tract infection, viral infection) requiring treatment in the 4 weeks prior to Visit 1, or an active respiratory infection at time of the Screening Visit.
5. Subject has a clinically significant abnormal finding on the physical examination, medical history, vital signs, ECG, lung x-ray or clinical laboratory results that could interfere with, or for which use of the study products might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study.
6. Subjects who have used any nicotine or tobacco product other than e-cigarettes or factory-made combustible cigarettes in the 14 days prior to the Visit 1.
7. Subjects who are self-reported or observed (during the trial session at Visit 2) non inhalers during ENDS/cigarette use.
8. Subjects who have used any prescription or over-the-counter (OTC) smoking cessation treatments, including, but not limited to any form of nicotine replacement therapy (NRT), varenicline, cytisine, or bupropion within 30 days prior to Visit 1.
9. Is planning to quit smoking during the study or postponing a quit attempt in order to participate in the study.
10. Subjects who have used prescription or OTC bronchodilator medication (e.g., inhaled or oral β adrenergic agonists, anticholinergics, glucocorticoids, cromones, or theophylline) to treat a chronic condition within the 12 months prior to Visit 1 or have a history of lung disease.
11. Subjects who have received any medications or substances that interfere with the cyclooxygenase pathway within 14 days prior to Visit 1 or are known to be strong inducers or inhibitors of cytochrome P450 (CYP) enzymes within 14 days or 5 half lives of the drug (whichever is longer) prior to Visit 1.
12. Women who are pregnant or who have a positive urine pregnancy test.
13. Women who are breast-feeding.
14. Subject has a history or diagnosis of adult asthma, COPD (including emphysema and chronic bronchitis), or use of an inhaler within the past 3 months.
15. Subject has been hospitalized in the 28 days prior to the Visit 1.
16. Subject has a history of schizophrenia, psychosis, or bipolar disorder.
17. Subject provides a positive drugs of abuse urine test at Visit 1. Tested drugs will include cocaine, amphetamines, methamphetamines, opiates (morphine, heroin), barbiturates, and benzodiazepine.
18. Subject has a self-reported use of more than 21 drinks per week. A drink is defined as 25 ml of spirits (e.g., whisky, vodka), 250 ml of beer, or 75 ml of wine.
19. Subjects who have lost or donated more than 450 mL of blood within the 2 months preceding the first product use.
20. Subject is an employee of the sponsor or the study site, or members of their immediate family.
21. In the opinion of the investigator, the subject should not participate in this study.
22. A history of allergy/oversensitivity to the ingredients of the study products.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-07-23 (Actual)

PRIMARY OUTCOMES:
Baseline-adjusted plasma nicotine Cmax0-120 | 0-120 minutes
  Maximum baseline-adjusted plasma concentration of nicotine from time zero to 120 minutes after the start of product use
Baseline-adjusted plasma nicotine Tmax0-120 | 0-120 minutes
  Baseline-adjusted plasma nicotine Tmax following defined product use
Baseline-adjusted plasma nicotine AUC0-120 | 0-120 minutes
  Baseline-adjusted area under the plasma nicotine concentration-versus-time curve from time zero to 120 minutes after the start of product use
Baseline-adjusted plasma nicotine Cmax0-180 | 0-180 minutes
  Maximum baseline-adjusted plasma concentration of nicotine from time zero to 180 minutes after the start of product use
Baseline-adjusted plasma nicotine Tmax0-180 | 0-180 minutes
  Baseline-adjusted plasma nicotine Tmax following both defined and ad libitum product use
Baseline-adjusted plasma nicotine AUC0-180 | 0-180 minutes
  Baseline-adjusted area under the plasma nicotine concentration-versus-time curve from time zero to 180 minutes after the start of product use
Product liking | 180 minutes
  Visual analog scale product liking assessment; scale from 0 to 100 with higher scores representing stronger liking.
Intent to Use Product Again | 180 minutes
  Visual analog scale intent to use product again assessment; scale from 0 to 100 with higher scores representing stronger intent to use the product again.
Urge to Smoke | 0-180 minutes
  Visual analog scale urge to smoke assessment; scale from 0 to 100 with higher scores representing stronger urge to smoke.
Product Evaluation Scale | 180 minutes
  Subjective effects assessment using Product Evaluation Scale, which included 21 items with responses recorded on a scale of 1 to 7 ranging from 'Not at all' to 'Extremely'.
Mass change | 0-5 minutes and 120-180 minutes
  Mass change in grams of ENDS products during use sessions

SECONDARY OUTCOMES:
Puff duration | 120-180 minutes
  Puff duration from puffing topography measurements
Puff volume | 120-180 minutes
  Puff volume from puffing topography measurements
Peak puff flow rate | 120-180 minutes
  Peak puff flow rate from puffing topography measurements
Average puff flow rate | 120-180 minutes
  Average puff flow rate from puffing topography measurements
Inter-puff interval | 120-180 minutes
  Time between puffs from puffing topography measurements

OTHER OUTCOMES:
Heart rate | 0-180 minutes
  Heart rate measurements made to assess safety
Blood pressure | 0-180 minutes
  Blood pressure measurements made to assess safety
Adverse events | From screening through study completion, an average of 1 month
  Adverse event reporting

CONTACTS AND LOCATIONS:
Overall Officials: Anna O Popko, MD, Principal Investigator — MTZ Clinical Research Sp z.o.o.
Locations (1):
- MTZ Clinical Research Sp. z o.o., Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fearon IM, Gilligan K, Seltzer RGN, McKinney W. A randomised, crossover, clinical study to assess nicotine pharmacokinetics and subjective effects of the BIDI(R) stick ENDS compared with combustible cigarettes and a comparator ENDS in adult smokers. Harm Reduct J. 2022 Jun 2;19(1):57. doi: 10.1186/s12954-022-00638-0. PMID 35655314